CLINICAL TRIAL: NCT04303507
Title: Chloroquine/ Hydroxychloroquine Prevention of Coronavirus Disease (COVID-19) in the Healthcare Setting; a Randomised, Placebo-controlled Prophylaxis Study (COPCOV)
Brief Title: Chloroquine/ Hydroxychloroquine Prevention of Coronavirus Disease (COVID-19) in the Healthcare Setting
Acronym: COPCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VIR20001
Record Dates: First submitted 2020-03-06; First posted 2020-03-11 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-05

CONDITIONS: COVID19; Coronavirus; Acute Respiratory Illnesses
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Chloroquine; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chloroquine or Hydroxychloroquine (Experimental): In Asia, the participant will receive chloroquine.
  In Europe, the participant will receive hydroxychloroquine
  Specific drug allocation will be determined by country prior to activation based upon factors such as inventory availability and importation requirements
  Interventions: Drug: Chloroquine or Hydroxychloroquine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chloroquine or Hydroxychloroquine — A loading dose of 10 mg base/ kg followed by 155 mg daily (250mg chloroquine phosphate salt or 200mg of or hydroxychloroquine sulphate) will be taken for 3 months
  Arms: Chloroquine or Hydroxychloroquine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study is a double-blind, randomised, placebo-controlled trial that will be conducted primarily in healthcare settings and other facilities directly involved in COVID-19 case management. We will recruit healthcare workers and other persons at risk of contracting COVID-19, who can be followed reliably for 5 months. The initial aim was to recruit 40,000 participants and we predict an average of 400-800 participants per site in 50-100 sites.

The participant will be randomised to receive either chloroquine or placebo (1:1 randomisation), or to hydroxychloroquine or placebo (1:1 randomisation). A loading dose of 10mg base/kg (four 155mg tablets for a 60kg subject), followed by 155 mg daily (250mg chloroquine phosphate salt/ 200mg hydroxychloroquine sulphate) will be taken for 3 months.

If the participant is diagnosed with COVID-19, they will take continue to take the study medication until:

* 90 days after enrolment (i.e., completion of kit)
* hospitalised due to COVID-19 disease (i.e., not for quarantine purposes) in which case they will stop, or
* advised to stop by their healthcare professional for other reasons

Episodes of symptomatic respiratory illness, including symptomatic COVID-19, and clinical outcomes will be recorded in the Case Record Form during the follow-up period.

This study is funded by Wellcome Trust Grant reference 221307/Z/20/Z.

ELIGIBILITY:
Study Participants The study population is adult healthcare workers and other persons defined by the site investigator at risk of contracting COVID-19.

Inclusion Criteria

1. Participant is willing and able to give informed consent for participation in the study and agrees with the study and its conduct
2. Agrees not to self-medicate with chloroquine, hydroxychloroquine or other potential antivirals
3. Adults (exact age is dependent on countries) less than 70 years old at the time of consent
4. Not previously diagnosed with COVID-19
5. Not currently symptomatic with an ARI
6. Participant is a healthcare worker or is a person at risk of contracting COVID-19.
7. Possesses an internet-enabled smartphone (Android or iOS)

Exclusion Criteria:

1. Hypersensitivity reaction to chloroquine, hydroxychloroquine or 4-aminoquinolines
2. Contraindication to taking chloroquine as prophylaxis e.g. known epileptic, known creatinine clearance < 10 ml/min
3. Already taking chloroquine, hydroxychloroquine or 4-aminoquinolines, or history of these medications within the previous 7 days
4. Taking prohibited medications
5. Known retinal disease
6. Inability to be followed up for the trial period
7. Known prolonged QT syndrome (however ECG is not required at baseline)
8. Known pregnancy or women who are actively trying to become pregnant
9. Prior diagnosis of porphyria
10. Previously received any dose of COVID-19 vaccine

The investigator may consult the physician's guidance documents for any further questions regarding eligibility of potential participants.

Prohibited medications for the purpose of study enrollment include:

* Antiarrhythmic medications: digoxin, amiodarone, sotalol, flecainide
* Antiparasitic/malarial agents: mefloquine, halofantrine, praziquantel
* Antibiotics: levofloxacin, moxifloxacin, ciprofloxacin, azithromycin, clarithromycin, erythromycin
* Antifungal drugs: fluconazole, ketoconazole, itraconazole, terfenadine
* Psychoactive drugs: lithium, quetiapine, chlorpromazine, thioridazine, ziprasidone, haloperidol, droperidol, methadone
* Migraine treatment: sumatriptan
* Antihistamines: astemizole
* Antiemetics: prochlorperazine, metoclopramide
* Cancer treatments: abiraterone, dabrafenib, dacomitinib, enzalutamide, idelalisib, mitotane
* Other specific drugs: ciclosporin, conivaptan, agalsidase alfa or beta, mifepristone, stiripentol

PrincipaI Investigators will also be directed to crediblemeds.org to check other agents that may prolong QT interval

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4652 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Number of symptomatic COVID-19 infections | Approximately 90 days
  Number of symptomatic COVID-19 infections will be compared between the chloroquine or hydroxychloroquine and placebo groups

SECONDARY OUTCOMES:
Symptoms severity of COVID-19 | Approximately 90 days
  Symptoms severity of COVID-19 will be compared between the two groups using a respiratory severity score.
Number of asymptomatic cases of COVID-19 | Approximately 90 days
  Number of asymptomatic cases of COVID-19 will be determined by comparing serology in all participants at time of enrolment and at the end of follow up.
Number of symptomatic acute respiratory illnesses | Approximately 90 days
  Number of symptomatic acute respiratory illnesses will be compared between the chloroquine or hydroxychloroquine and placebo groups.
Severity of symptomatic acute respiratory illnesses | Approximately 90 days
  Severity of symptomatic acute respiratory illnesses will be compared between the chloroquine or hydroxychloroquine and placebo groups.

OTHER OUTCOMES:
Genetic loci and levels of biochemical components will be correlated with frequency of COVID-19, ARI and disease severity. | Approximately 90 days
  Genetic loci and levels of biochemical components will be correlated with frequency of COVID-19, Acute Respiratory Infection and disease severity.
Assess the impact of chloroquine or hydroxychloroquine prophylaxis on number of days lost to work during the pandemic. | Approximately 90 days
  Number of days lost to work in relation to the treatment arm
Assess the impact of chloroquine or hydroxychloroquine prophylaxis on healthcare costs | Approximately 90 days
  The trial will collect data on monetary costs associated with the use of healthcare resources and determine the effects between treatment groups.
Assess the impact of chloroquine or hydroxychloroquine prophylaxis on quality of life measures using the quality of life questionnaire (EQ-5D-3L) | Approximately 90 days
  The trial will collect data on health-related quality of life using the quality of life questionnaire (EQ-5D-3L) to determine the effects between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: William Schilling, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (25):
- Benin (2):
  - Centre Hospitalier et Universitaire de Zone Abomey-Calavi, Abomey-Calavi
  - Hospital De Zone Allada, Allada
- Côte d’Ivoire (2):
  - University Hospital Center of Angre, Abidjan
  - University Hospital Center of Bouake, Bouaké
- Indonesia (5):
  - Airlangga University Hospital (UNAIR), Surabaya, East Java
  - Husada Utama Hospital, Surabaya, East Java
  - Bunda Thamrin Hospital, Medan, North Sumatra
  - Murni Teguh Memorial Hospital, Medan, North Sumatra
  - Sardjito Hospital, Yogyakarta
- Kenya (2):
  - Fountain Healthcare Hospital, Eldoret
  - Mbagathi County Hospital, Nairobi
- Mali (2):
  - The Bamako Hospital of Dermatology, Bamako
  - Hospital Of Mali, Bamako
- B.P. Koirala Institute of Health Sciences, Dharān, Nepal
- The Aga Khan University Hospital, Karachi, Pakistan
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand
- United Kingdom (8):
  - University Hospitals Of Morecambe Bay NHS Foundation Trust, Kendal, Cumbria
  - The Dudley Group NHS Foundation Trust, Dudley, West Midlands
  - Birmingham & Solihull Mental Health NHS Trust, Birmingham
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Rotherham, Doncaster And South Humber NHS Foundation Trust, Doncaster
  - Imperial College Healthcare NHS Trust, London
  - Oxford University Hospital NHS Foundation Trust, Oxford
- Zambart, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, suitably anonymised clinical data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with other researchers to use in the future.
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing

REFERENCES:
- [Derived] Winters J, Schilling WH. Approval delays in multi-country COVID-19 trials: the case of COPCOV and the risk of therapeutic inertia. Trials. 2025 Dec 16:10.1186/s13063-025-09300-z. doi: 10.1186/s13063-025-09300-z. Online ahead of print. PMID 41402852
- [Derived] Schilling WHK, Mukaka M, Callery JJ, Llewelyn MJ, Cruz CV, Dhorda M, Ngernseng T, Waithira N, Ekkapongpisit M, Watson JA, Chandna A, Nelwan EJ, Hamers RL, Etyang A, Beg MA, Sow S, Yavo W, Allabi AC, Basnyat B, Sharma SK, Amofa-Sekyi M, Yonga P, Adler A, Yuentrakul P, Cope T, Thaipadungpanit J, Rienpradub P, Imwong M, Abdad MY, Blacksell SD, Tarning J, Goudjo FF, Dossou AD, Konate-Toure A, Assi SB, Ouffoue K, Nasronudin N, Rachman BE, Romadhon PZ, Dewanto DD, Heryana MO, Novi T, Pasaribu AP, Mutiara M, Nasution MPR, Khairunnisa K, Dalimunthe FA, Airlangga E, Fahrezzy A, Subronto Y, Ananda NR, Rahardjani M, Rimainar A, Lucinde RK, Timbwa M, Onyango OE, Agutu C, Akech S, Hamaluba M, Kipyego J, Ngachi O, Haidara FC, Traore OY, Diarra F, Khanal B, Dahal P, Shrestha S, Rijal S, Kabore Y, Adehossi E, Guindo O, Qamar FN, Kazi AM, Woodrow CJ, Laird S, Cheeba M, Ayles H, Cheah PY, Taylor WRJ, Batty EM, Chotivanich K, Pukrittayakamee S, Phumratanaprapin W, von Seidlein L, Dondorp A, Day NPJ, White NJ; COPCOV Collaborative Group. Evaluation of hydroxychloroquine or chloroquine for the prevention of COVID-19 (COPCOV): A double-blind, randomised, placebo-controlled trial. PLoS Med. 2024 Sep 12;21(9):e1004428. doi: 10.1371/journal.pmed.1004428. eCollection 2024 Sep. PMID 39264960
- [Derived] Kabore Y, Vatrinet R, Guindo O, Moussa SH, Schilling WHK, Grais RF. Reflections on Participation in a Trial on Hydroxychloroquine as Prevention for COVID-19 among Health Workers in Niger. Am J Trop Med Hyg. 2023 Aug 14;109(3):511-514. doi: 10.4269/ajtmh.22-0606. Print 2023 Sep 6. PMID 37580026
- [Derived] Akhtar S, Das JK, Ismail T, Wahid M, Saeed W, Bhutta ZA. Nutritional perspectives for the prevention and mitigation of COVID-19. Nutr Rev. 2021 Feb 11;79(3):289-300. doi: 10.1093/nutrit/nuaa063. PMID 33570583
- See also: Related Info — https://www.tropmedres.ac/covid-19/copcov

DOCUMENTS (2):
  • Study Protocol (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT04303507/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT04303507/SAP_001.pdf